CLINICAL TRIAL: NCT07161648
Title: Use of Neuromuscular Electrical Stimulation to Prevent Exercise Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Christopher Bell, Associate Prof, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5208
Record Dates: First submitted 2025-09-02; First posted 2025-09-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Fat Metabolism
Keywords: exercise; exercise resistance; electrical stimulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Establishing the normal benefit of exercise (No Intervention): Study participants will complete treadmill exercise. During the same day, they will walk a minimum of 8,500 steps. The next day, fat oxidation will be measured after eating a high-fat meal.
- Demonstrating exercise resistance (No Intervention): Study participants will complete treadmill exercise. They will walk no more than 5,000 steps on the same day. The next day, fat oxidation will be measured after eating a high-fat meal.
- Trying to prevent exercise resistance (Experimental): Study participants will complete treadmill exercise. They will walk no more than 5,000 steps on the same day. They will receive 100 minutes of neuromuscular electrical stimulation. The next day, fat oxidation will be measured after eating a high-fat meal.
  Interventions: Other: neuromuscular electrical stimulation

INTERVENTIONS:
Other: neuromuscular electrical stimulation — The study participants will engage in 100-minutes of neuromuscular electrical stimulation (NMES). NMES pads are sticky pieces of plastic, similar in size to a 25-cent coin. The pads will be placed on the bellies of thigh muscles (the vastus lateralis, vastus medialis), and calf muscles (the long and short head of the gastrocnemius). These skeletal muscles are selected due to their size (thereby promoting a bigger increase for metabolic rate compared with a small muscle), because they are relatively superficial, and because previous published studies of NMES used these anatomical locations.
  Arms: Trying to prevent exercise resistance

SUMMARY:
The study will find out if 100 minutes of electrical stimulation of muscle prevents the unfavorable consequence of insufficient exercise.

DETAILED DESCRIPTION:
Exercise resistance is characterized by the absence of exercise induced improvements in fat metabolism following a meal, and results from prolonged sedentary behavior between successive workouts (i.e. 2+ sedentary days between exercise bouts). The suggested energy expenditure threshold for avoiding exercise resistance is the equivalent of walking ~8,500 steps/day. However, population data indicate that the typical adult in the US only walks 5,000 steps/day (i.e. 3,500 steps below the threshold). Neuromuscular Electrical Stimulation (NMES) evokes skeletal muscle contractions and increases energy expenditure. The hypothesis to be explored in this current proposal is: NMES will prevent exercise resistance. The plan is to induce exercise resistance via short-term abstention from activity other than exercise, and then on a separate occasion, use NMES to prevent exercise resistance (i.e. the short-term abstention from exercise will be "replaced" with NMES).

ELIGIBILITY:
Inclusion Criteria:

* Regularly active (more than 30 minutes of exercise per day, 3 days per week, over the previous 12 months)
* Ability to complete at least one hour of treadmill exercise (i.e. jogging/running),
* Willing to abstain from caffeine and alcohol for 24-hours prior to three different study visits
* Competency in English

Exclusion Criteria:

* Current or previous injuries that may hinder a participant's ability to exercise on a treadmill
* A history of cardiopulmonary disorder that may be contra-indicative to treadmill exercise
* Current use of cardio-pulmonary medication to treat a cardio-pulmonary condition
* Currently breastfeeding
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fat oxidation | Blood will be sampled and triglyceride concentration measured. Study participants will eat a meal. Blood will be sampled and triglyceride concentration measured every 30-minutes for 4 hours.
  Circulating triglyceride concentration after eating a high fat meal.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Group descriptive statistics (e.g. average and standard deviation) will be shared.